CLINICAL TRIAL: NCT05279144
Title: Comparison of Intramuscular Injection From Two Different Sites in Children Pain and Fear: A Randomized Controlled Study
Brief Title: Comparison of Intramuscular Injection From Two Different Sites in Children
Acronym: Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Dr, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ÖZNUR TİRYAKİ
Record Dates: First submitted 2022-02-02; First posted 2022-03-15 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Application Site Infection
Keywords: children; fear; pain; Intramuscular injection; injection site
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Comparison of vastus lateralis (VL) and ventrogluteal (VG) region applications in terms of pain and fear in safe and evidence-based intramuscular injection application in children.
Masking Description: It is known by the researcher which group the participants belong to. 1 week VL, 1 week VG application will be done.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ventrogluteal region IM injection will be applied to the children in the intervention group, which is recommended by the literatureIn order to ensure that the children in the groups are similar in terms of two factors (same drug, same nurse) in the assignment, they will be assigned to the groups first by stratified sampling method and then by simple random sampling (http://www1.assumption.edu/users/avadum/applets/RandAssin/Groupgen). .html). In the case of a 5% margin of error and an effect width of 0.70 at 80% power, the total number of patients, including 40 control and 40 intervention groups, who met the inclusion criteria of the study, was determined as 80.
  Interventions: Other: Ventroguleal
- No Intervention (No Intervention): Vastus Lateralis IM injection, which is the routine practice of the clinic, will be applied to the children in the control group of the study. In order to ensure that the children in the groups are similar in terms of two factors (same drug, same nurse) in the assignment, they will be assigned to the groups first by stratified sampling method and then by simple random sampling (http://www1.assumption.edu/users/avadum/applets/RandAssin/Groupgen). .html). In the case of a 5% margin of error and an effect width of 0.70 at 80% power, the total number of patients, including 40 control and 40 intervention groups, who met the inclusion criteria of the study, was determined as 80.

INTERVENTIONS:
Other: Ventroguleal — Vastus Lateralis
  Other Names: Control
  Arms: Experimental

SUMMARY:
Administration of intramuscular injections (IM) is now common practice in pediatric clinical settings. For this reason, nurses should both update their clinical skills and provide evidence-based practices to children. The aim of this study; The aim of this study is to compare vastus lateralis (VL) and ventrogluteal (VG) region applications in terms of pain and fear in safe and evidence-based intramuscular injection application in children.

H0: There is no difference in terms of pain and fear between the children aged 4-6 years who received IM from the vastus lateralis (VL) region and those who received IM from the ventrogluteal (VG) region.

H1: Children between the ages of 4 and 6 years IM administered from the vastus lateralis (VL) region have higher pain than those administered IM from the ventrogluteal (VG) region.

H2: The fear of children aged 4-6 years who underwent IM from the vastus lateralis (VL) region is higher than that of children who were administered IM from the Ventrogluteal (VG) region.

DETAILED DESCRIPTION:
Intramuscular injection (IMI) is widely used in the pediatric emergency department and is a cause of pain for children. The aim of this study is to compare the vastus lateralis (VL) and ventrogluteal (VG) region applications in terms of pain and fear in intramuscular injection application in children aged 4-6 years.

The population of the study consists of children aged 4-6 years who applied to the emergency department for IM injection. The sample of the study consisted of 80 children (40 in the intervention group, 40 in the control group) who met the inclusion criteria within the specified date range.

The injection technique was explained to the parents and children by showing the location of the VL and VG regions on the model doll. Both parents and their children were informed about the research. Written and verbal consent was obtained from the parents and verbal consent was obtained from the children. It was decided to meet the control group for one week and the intervention group for one week in order to avoid any interference between the two groups. In which week the children will be included in which group was randomly determined in the computer environment. There are two stretchers and a privacy curtain between them in the injection room in the Pediatric Emergency Clinic where the research was conducted. The nurse in charge of the daily injection room changes. For each patient who comes for injection, the ordered prescription is checked first, and then it is entered into the hospital system. The ordered drug is based on 10 correct drug administration principles (1. Correct drug, 2. Correct dose, 3. Correct patient, 4. Correct time, 5. Correct route of administration, 6. Correct patient education, 7. Correct registration, 8. Confirmation of rejection. , 9. Correct drug preparation (form), 10. Correct answer). In order to determine whether a drug-related reaction has developed or not, the patient is observed until 15-30 minutes after the application (the time varies according to the drug). In the clinic, IM injection to children aged 4-6 years is routinely performed by nurses from the VL region.

Data collection instruments Questionnaire form, Wong-baker faces pain rating scale (WBFPTS), Children's Fear Scale (CFS) were used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age group of 4-6
* Ordering Prendol amp IM by the doctor,
* IM application in pediatric emergency,
* Absence of a disease that causes chronic pain,
* Absence of a neurodevelopmental disorder,
* Not taking analgesics in the last 6 hours,
* No history of fainting during the injection,
* Absence of mental retardation,
* Absence of scar tissue or muscle atrophy in the area to be injected,
* Being in the 10th to 90th percentile
* Families and children agree to participate in the research.

Exclusion Criteria:

* - being less than 4 years old,
* Over 6 years of age,
* Scar or muscle atrophy at the injection site,
* The child or parent has communication problems,
* The percentile is below 10 (cachectic) or over 90 (obese),
* Families and children do not agree to participate in the research.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
children pain | through study completion, an average of 3month
  Comparison of VL and VG injection application in terms of pain in children aged 4-6 years.
  Wong-baker faces pain rating scale (Wong-baker) It can be applied between the ages of 3-18. It can be applied in many pains such as acute, chronic and postoperative pain. It was developed by Wong and Baker. The horizontal plane also contains six hand-drawn facial expressions. It is scored between 0-10 points. It symbolizes the phrase "no pain" with a smiley face on the far left. Pain increases from sodan to right. On the far right, there is a crying facial expression with tears representing the expression "unbearable pain".
fear | through study completion, an average of 3month
  Comparison of VL and VG injection application in terms of fear in children aged 4-6 years.
  Children's Fear Scale CFS is used to scale the child's anxiety level. The CDS is a scale from 0-4, consisting of showing five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK MENEKŞE, Assis prof., Study Director — Sakarya University; NURSAN ÇINAR, Proffesor, Principal Investigator — Sakarya University; BAHRİ ELMAS, Assoc Prof, Principal Investigator — Sakarya University; ÖNER ÖZDEMİR, Proffesor, Principal Investigator — Sakarya University
Locations (1):
- Sakarya Education and Training Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No